CLINICAL TRIAL: NCT04700163
Title: A Phase 1, Open Label, Dose-escalation Study of the Safety and Pharmacokinetics of a Combination of Two Anti-SARS-CoV-2 mAbs (C144-LS and C135-LS) in Healthy Volunteers
Brief Title: RU Anti-SARS-CoV-2 (COVID-19) mAbs in Healthy Volunteers
Acronym: RU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RUCOV1; CGA-1015 (Other: Rockefeller University IRB)
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Covid19
Keywords: Monoclonal antibody; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — ogalvibart, crexavibart drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- S1 - low dose (Experimental): 100 mg of C144-LS and 100 mg of C135-LS, subcutaneously
  Interventions: Biological: C144-LS and C-135-LS
- S2 - mid dose (Experimental): 200 mg of C144-LS and 200 mg of C135-LS, subcutaneously
  Interventions: Biological: C144-LS and C-135-LS
- V1 - low dose (Experimental): 1.5 mg/kg of C144-LS and 1.5 mg/kg of C135-LS, intravenously
  Interventions: Biological: C144-LS and C-135-LS
- V2 - mid dose (Experimental): 5 mg/kg of C144-LS and 5 mg/kg of C135-LS, intravenously
  Interventions: Biological: C144-LS and C-135-LS
- V3 - high dose (Experimental): 15 mg/kg of C144-LS and 15 mg/kg of C135-LS, intravenously
  Interventions: Biological: C144-LS and C-135-LS

INTERVENTIONS:
Biological: C144-LS and C-135-LS — A combination of two highly neutralizing anti-SARS-CoV-2 mAbs targeting two distinct epitopes on the receptor protein binding domain (RBD) of the SARS-CoV-2 spike protein

SUMMARY:
This is a first-in-human, open label, single dose, dose-escalation phase 1 study to evaluate the safety and pharmacokinetics of a combination of two highly neutralizing anti-SARS-CoV-2 mAbs targeting two distinct epitopes on the receptor protein binding domain (RBD) of the SARS-CoV-2 spike protein in healthy volunteers.

DETAILED DESCRIPTION:
The study has a standard 3+3 phase 1 dose escalation design. Study participants will receive subcutaneous injections of C144-LS and C135-LS at 4ml (approximately 100mg of each antibody administered separately) or 8ml (approximately 200mg of each antibody administered separately), or sequential intravenous infusions of C144-LS and C135-LS, at one of three increasing dose levels (1.5 mg/kg, 5 mg/kg and 15 mg/kg of each antibody).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use one effective method of contraception from 10 days prior to the antibody administration until 6 months after investigational product (IP) administration.

Exclusion Criteria:

* Weight > 110 kg for groups S1 and S2 only
* History of prior positive SARS-CoV-2 RT-PCR or SARS-CoV-2 serology.
* Active respiratory or non-respiratory symptoms consistent with COVID-19.
* Medically attended acute illness or hospitalization (ie, >24 hours) for any reason within 30 days prior to screening.
* Acute exacerbation of a chronic pulmonary condition (eg, chronic obstructive pulmonary disease [COPD], asthma exacerbations, or uncontrolled hypertension, as defined by a systolic blood pressure > 180 and/or diastolic blood pressure > 120, in the presence or absence of anti-hypertensive medications) in the past 6 months prior to screening.
* Use of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
* Other clinically significant acute or chronic medical condition that in the opinion of the investigator would preclude participation.
* Laboratory abnormalities in the parameters listed:

  * Absolute neutrophil count less than 1,500 K/mcL;
  * Hemoglobin less than 10.5 gm/dL if female; less than 11 gm/dL if male;
  * Platelet count less than 125,000 K/mcL;
  * ALT less than 1.25 x ULN; AST less than 1.25 x ULN;
  * Total bilirubin less than 1.25 x ULN;
  * Creatinine less than 1.1 x ULN;
* Pregnancy or lactation.
* Any vaccination within 14 days prior to SARS-CoV-2 mAbs administration (except influenza vaccine).
* History of prior receipt of any SARS-CoV-2 vaccine or antibodies, including convalescent plasma.
* Known allergy/sensitivity or any hypersensitivity to components of the investigational agents.
* History of severe reaction to a vaccine or monoclonal antibody administration or history of severe allergic reactions.
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gaebler, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schafer A, Muecksch F, Lorenzi JCC, Leist SR, Cipolla M, Bournazos S, Schmidt F, Maison RM, Gazumyan A, Martinez DR, Baric RS, Robbiani DF, Hatziioannou T, Ravetch JV, Bieniasz PD, Bowen RA, Nussenzweig MC, Sheahan TP. Antibody potency, effector function, and combinations in protection and therapy for SARS-CoV-2 infection in vivo. J Exp Med. 2021 Mar 1;218(3):e20201993. doi: 10.1084/jem.20201993. PMID 33211088
- [Background] Weisblum Y, Schmidt F, Zhang F, DaSilva J, Poston D, Lorenzi JC, Muecksch F, Rutkowska M, Hoffmann HH, Michailidis E, Gaebler C, Agudelo M, Cho A, Wang Z, Gazumyan A, Cipolla M, Luchsinger L, Hillyer CD, Caskey M, Robbiani DF, Rice CM, Nussenzweig MC, Hatziioannou T, Bieniasz PD. Escape from neutralizing antibodies by SARS-CoV-2 spike protein variants. Elife. 2020 Oct 28;9:e61312. doi: 10.7554/eLife.61312. PMID 33112236
- [Background] Barnes CO, Jette CA, Abernathy ME, Dam KA, Esswein SR, Gristick HB, Malyutin AG, Sharaf NG, Huey-Tubman KE, Lee YE, Robbiani DF, Nussenzweig MC, West AP Jr, Bjorkman PJ. SARS-CoV-2 neutralizing antibody structures inform therapeutic strategies. Nature. 2020 Dec;588(7839):682-687. doi: 10.1038/s41586-020-2852-1. Epub 2020 Oct 12. PMID 33045718
- [Result] Robbiani DF, Gaebler C, Muecksch F, Lorenzi JCC, Wang Z, Cho A, Agudelo M, Barnes CO, Gazumyan A, Finkin S, Hagglof T, Oliveira TY, Viant C, Hurley A, Hoffmann HH, Millard KG, Kost RG, Cipolla M, Gordon K, Bianchini F, Chen ST, Ramos V, Patel R, Dizon J, Shimeliovich I, Mendoza P, Hartweger H, Nogueira L, Pack M, Horowitz J, Schmidt F, Weisblum Y, Michailidis E, Ashbrook AW, Waltari E, Pak JE, Huey-Tubman KE, Koranda N, Hoffman PR, West AP Jr, Rice CM, Hatziioannou T, Bjorkman PJ, Bieniasz PD, Caskey M, Nussenzweig MC. Convergent antibody responses to SARS-CoV-2 in convalescent individuals. Nature. 2020 Aug;584(7821):437-442. doi: 10.1038/s41586-020-2456-9. Epub 2020 Jun 18. PMID 32555388
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened for participation and screened out if did not meet eligibility criteria.
  Participants enrolled sequentially in the study, following a dose escalation scheme as per protocol.
Groups:
- S3 - Open Label: 200 mg of C144-LS and 200 mg of C135-LS or placebo, subcutaneously.
  C144-LS and C-135-LS: A combination of two highly neutralizing anti-SARS-CoV-2 mAbs targeting two distinct epitopes on the receptor protein binding domain (RBD) of the SARS-CoV-2 spike protein
Period: Overall Study
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Started | 3 | 3 | 3 | 3 | 3 | 8
Completed | 3 | 3 | 3 | 3 | 3 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- S3 - Open Label: 200 mg of C144-LS and 200 mg of C135-LS or placebo, subcutaneously
  C144-LS and C-135-LS: A combination of two highly neutralizing anti-SARS-CoV-2 mAbs targeting two distinct epitopes on the receptor protein binding domain (RBD
- Total: Total of all reporting groups
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 3 | 8 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42 [28 to 58] | 39 [33 to 47] | 39 [26 to 58] | 52 [51 to 54] | 54 [38 to 64] | 38 [24 to 59] | 44 [24 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 0 | 0 | 3 | 6
  Male | 3 | 2 | 1 | 3 | 3 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 1 | 1 | 4
  Not Hispanic or Latino | 3 | 2 | 2 | 3 | 2 | 7 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 0 | 1 | 3 | 8
  White | 0 | 2 | 2 | 2 | 1 | 2 | 9
  More than one race | 1 | 0 | 0 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Grade 2 and Higher Adverse Events 4 Weeks After Administration.
Description: The number of participants with treatment-related solicited and unsolicited grade 2 adverse events (including confirmed laboratory abnormalities).
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Grade 3 and Higher Adverse Events 4 Weeks After Administration.
Description: The number of participants with treatment-related solicited and unsolicited grade 3 adverse events (including confirmed laboratory abnormalities).
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Related Serious Adverse Events (SAEs) Throughout the Study Period
Description: The number of participants with treatment-related solicited serious adverse events.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Elimination Half-life (t1/2) of C135-LS and C144-LS
Description: Half-life of C135-LS and C144-LS when administered intravenously or subcutaneously in healthy volunteers
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7
days
  C135-LS Half-life | 79.85 (10.84) | 89.55 (17.06) | 90.79 (15.11) | 91.91 (12.57) | 96.24 (13.56) | 89.55 (17.06)
  C144-LS Half-life | 80.96 (14.58) | 107.3 (29.21) | 96.37 (11.48) | 114.4 (3.444) | 103.5 (14.10) | 107.3 (29.2)

5. Primary Outcome: Clearance Rate of C135-LS and C144-LS
Description: Clearance rate of C135-LS and C144-LS when administered intravenously or subcutaneously in healthy volunteers
Time Frame: 48 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ml/day
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6
ml/day
  C135-LS Clearance | 75.34 (33.54) | 70.58 (22.81) | 53.13 (19.61) | 70.88 (13.89) | 62.75 (19.56) | 70.58 (22.81)
  C144-LS Clearance | 61.54 (7.105) | 61.43 (16.70) | 35.34 (26.85) | 50.96 (7.965) | 44.86 (6.584) | 61.43 (16.70)

6. Primary Outcome: Area Under the Curve of C135-LS and C144-LS
Description: Area under the curve of C135-LS and C144-LS when administered intravenously or subcutaneously in healthy volunteers
Time Frame: 48 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (micrograms x day)/ml
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6
(micrograms x day)/ml
  C135-LS AUC | 1327 (33.54) | 2833 (22.81) | 1873 (6.6) | 6213 (27.92) | 19626 (6.464) | 2833 (22.81)
  C144-LS AUC | 1625 (35.03) | 3256 (16.79) | 2816 (13.42) | 8641 (31.4) | 27452 (3.205) | 3256 (16.79)

7. Secondary Outcome: Investigational Product (IP)-Related Adverse Events During Study Follow up.
Description: The number of participants with treatment-related adverse events
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 8
Participants | 0 | 1 | 0 | 0 | 2 | 0

8. Secondary Outcome: Anti-C144-LS and Anti-C135-LS Antibodies in All Study Groups.
Description: Proportion of individuals with treatment-induced anti-drug antibodies against each mAb and magnitude of the response
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6
Participants
  C135-LS ADA | 1 | 2 | 0 | 1 | 0 | 0
  C144-LS ADA | 1 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Definitions are the definitions from clinicaltrials.gov
Arm/Group | S1 - Low Dose | S2 - Mid Dose | V1 - Low Dose | V2 - Mid Dose | V3 - High Dose | S3 - Open Label
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/8
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/3 | 1/3 | 2/3 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S1 - Low Dose (N=3) | S2 - Mid Dose (N=3) | V1 - Low Dose (N=3) | V2 - Mid Dose (N=3) | V3 - High Dose (N=3) | S3 - Open Label (N=8)
Tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased blood glucose (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 Antibody Positive (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT04700163/Prot_SAP_000.pdf